CLINICAL TRIAL: NCT03221699
Title: Effects of a Zinc Oxide Underarm Formula on Normal and Injured Skin: A Randomized and Double-blind Trial in Healthy Volunteers
Brief Title: Effects of a Zinc Oxide Underarm Formula on Normal and Injured Skin in Healthy Volunteers
Acronym: ZINC-ON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lars Nannestad Jorgensen (Other)
Collaborators: Colgate Palmolive (Industry)
Responsible Party: Sponsor-Investigator, Lars Nannestad Jorgensen, Professor, MD, DrMedSci, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-16045754
Record Dates: First submitted 2017-03-30; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Microbiome of the Axillae
MeSH Terms: interventions — Food, Formulated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Placebo Comparator): Formula without ZnO
  Interventions: Other: Formula without ZnO
- intervention (Active Comparator): Formula with ZnO
  Interventions: Other: Formula with ZnO

INTERVENTIONS:
Other: Formula with ZnO — Forearms and axillae are treated by the volunteers once daily with a standardized amount of the roll-on with ZnO
  Arms: intervention
Other: Formula without ZnO — Forearms and axillae are treated by the volunteers once daily with a standardized amount of the roll-on without ZnO
  Arms: control

SUMMARY:
Bothersome odor from the axilla is in most cases caused by Corynebacterium spp. Anti-microbial effects of zinc oxide (ZnO) are well documented.

The overall objective of this study is to verify that repeated applications of a ZnO containing formulation can be directly linked to reduced growth of Corynebacterium spp. in the axillae.

DETAILED DESCRIPTION:
In the trial the effects of the ZnO formulation on the skin of the forearms and axillae are investigated simultaneously. In both locations the skin is treated daily with the ZnO/placebo formulations.

At day -8 skin areas of the forearms and the axillae are sampled by adhesive tape that is extracted in phosphate-buffered saline (PBS) and PBS extract analyzed on total proteins (BCA) and IL-1α. In the axillae swabs are taken for Corynebacterium spp. semi quantification and pH is measured in the axillae and on the forearm.

At day 0 treated skin areas of the forearms and the axillae are sampled by adhesive tape that is extracted in PBS and PBS extract analyzed on total proteins (BCA) and IL-1α, and compared to adjacent non-treated skin. In the axillae and on the forearms, swabs are first taken for Corynebacterium spp. semi quantification followed by wounding using ablative fractional (10%) carbon dioxide laser at 20 millijoule/microbeam and pediatric lancet. pH is measured in the axillae and on the forearm.

Progress of wound healing is assessed by dermatoscopy at days 3, 4 and 5. At day 5 swabs are taken in the axillae for Corynebacterium spp. semi quantification and pH is measured. Furthermore, skin areas of the axillae are sampled by adhesive tape that is extracted in PBS and PBS extract analyzed on total proteins (BCA) and IL-1α.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Age between 18 and 65 years
* Non-smoking
* Written informed consent

Exclusion Criteria:

* No current or past skin disorder
* Immunosuppressive treatment
* Pregnant and breast feeding women
* Hypersensitivity to zinc and/or other ingredients in the products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Growth of Corynebacterium spp. after 8 days of treatment | Day 0
  Skin surface swabs are cultured, and Corynebacterium spp. identified by light microscopy/MALDI-TOF mass spectrometry and semiquantified.

SECONDARY OUTCOMES:
Wound healing | Day 3, day 4 and day 5
  Dermatoscopy is used to assess the erythema, crust formation and healing
Quantification of total proteins and interleukin (IL)-1α | Day -8, day 0 and day 5
  Corneocytes are sampled on both forearms and axillae by adhesive tape (Sebutape®; CuDerm, Dallas, Texas, USA) for quantification of total proteins (BCA) and IL-1α levels by ELISA.
Changes in skin acidity level (pH) | Day -8 and day 5
  pH measurements are performed on both axillae
Pain | Day -8, day 0, day 3, day 4 and day 5
  McGill pain questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lars N Joergensen, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: No